CLINICAL TRIAL: NCT07273708
Title: Identification of an Immune Single Cell Transcriptomic Profile of Responder and Non-responder Hepatocellular Carcinoma Patients Treated With Immune-checkpoint Inhibitors
Acronym: HCC RNA-seq
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Salvatore Corallo, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 0014773/25
Record Dates: First submitted 2025-09-22; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Advanced HCC Treated by Systemic Immunotherapy
Keywords: HCC Organoids; HCC PBMCs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: Patients treated withi immune-check point inhibitor-based combinations as first-line treatment for advanced HCC

SUMMARY:
The study aims to analyze blood samples from patients with advanced hepatocellular carcinoma who are receiving systemic treatment with immunotherapy. The objective is to determine whether treatment exposure leads to changes in the transcriptomic patterns of peripheral blood mononuclear cells (PBMCs), if these changes are associated with treatment response, and whether certain pre-treatment transcriptomic signatures can predict response to treatment.

As an exploratory objective, PBMCs derived from patients exposed to immune checkpoint inhibitors will be co-cultured with their paired tumor cells in organoid cultures. This aims to assess whether these preclinical 3D models correlate with clinical outcomes.

DETAILED DESCRIPTION:
The primary pivotal objective of the study is to analyse the single cell transcriptome of peripheral blood mononuclear cells (PBMCs) in patients with HCC treated with immunotherapy to define if treatment exposure determines transcriptomic pattern changes and if some of these changes are associated with treatment response.

The secondary objective of the study is to investigate if some pre-treatment transcriptome signature of PBMCs is predictive of response and long-lasting response to treatment.

As an exploratory objective, the study investigators will analyse the interaction between patients' peripheral immune cells previously exposed to immune check-point inhibitors and their paired tumour cells in the organoid cultures.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of advanced HCC treated with atezolizumab plus bevacizumab or tremelimumab single dose plus durvalumab (STRIDE regimen) as first-line treament
2. age ≥18 and <90 years at time of signing informed consent
3. Signed Informed Consent Form

Exclusion Criteria:

1. Life expectancy of <12 months due to concomitant diseases
2. Active or history of autoimmune disease or immune deficiency on inflammatory chronic diseases
3. Ongoing drug abuse
4. History of malignancy other than HCC within 3 years prior to study entry with the following exception:

   1. Completely resected malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate 90%) and without evidence of recurrence for > 3 years prior to study entry
   2. adequately treated non-melanoma skin carcinoma or lentigo maligna without evidence of metastases.
   3. adequately treated carcinoma in situ of the cervix without evidence of recurrence
   4. localised prostate cancer
   5. adequately treated non invasive or in situ urothelial cancers
5. evidence or history of positive HIV test
6. inability to comply with the study protocol, in the investigator's judgment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with atezolizumab plus bevacizumab or tremelimumab single dose plus durvalumab (STRIDE regimen) as first-line treament for advanced HCC
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Analysis of the single cell profiling of peripheral blood mononuclear cells in patients with HCC treated with immunotherapy pre-therapy (T0) and the 3 months post-therapy (T3) to define if a difference between the two time points exists. | From enrollment untill 3 months after treatment start, (up to 120 days from study inclusion)
  The single cell profiling of peripheral blood mononuclear cells in patients with HCC treated with immunotherapy will be analised at two type points: before starting therapy(T0), and the 3 months post-therapy (T3). The difference of single cell profiling of the two paired time-points will be analysed.

SECONDARY OUTCOMES:
Correlation between transcriptome signature at baseline and treatment outcomes. | From enrollment to the time of best response to treatment, up to 24 months from enrollement
  To define if there is a correlation between baseline transcriptome signatures and treatment outcomes (duration of response, median progression-free survival, median overall survival)
Correlation between baseline gene clusters and treatment responses | From enrollment to the time of best response, up to 24 months from enrollment
  To identify baseline gene clusters that correlats with higher respose rates

OTHER OUTCOMES:
Exploring the interacton between PBMCs and tumor tissue in 3D culture system. | From enrollment untill 3 months after treatment start, (up to 120 days from study inclusion)
  To compare the percentage of apoptosis in tumor cells from patient-derived 3D culture systems of HCC, co-cultured with PBMC harvested after treatment with immune checkpoint inhibitors (ICIs), versus those co-cultured with baseline PBMCs collected at T0.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Pending privacy protection evaluation